CLINICAL TRIAL: NCT02083276
Title: Mecillinam for Treatment of Genital Chlamydia Infection in Asymptomatic Men
Brief Title: Mecillinam for Treatment of Genital Chlamydia Infection
Acronym: MecillinamCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment failure on study medication observed
Sponsor: Oslo University Hospital (Other)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Principal Investigator, Anne Olaug Olsen, MD PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1917; 2013-002379-17 (EudraCT Number)
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Chlamydia Trachomatis Infection; Chlamydial Urethritis
Keywords: Chlamydia trachomatis; Urethritis; Genital Diseases, Male
MeSH Terms: conditions — Urethritis; Genital Diseases, Male | interventions — Amdinocillin Pivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pivmecillinamhydrochlorid (Experimental): Selexid 400 mg x 3 , 7 days
  Interventions: Drug: Pivmecillinamhydrochlorid

INTERVENTIONS:
Drug: Pivmecillinamhydrochlorid — PO 400 mg x3 for 7 days
  Other Names: Selexid

SUMMARY:
The mainstay of treating both symptomatic and asymptomatic genital Chlamydia trachomatis infection has been macrolide antibiotics in the form of azithromycin, and alternatively tetracycline antibiotics in the form of doxycycline. Studies from the late nineties found a single dose of 1 g azithromycin to be equally effective as a 7 day course of 200 mg doxycycline a day. However, recent studies have reported increasing treatment failure that may indicate that resistance to macrolide antibiotics among Chlamydia trachomatis is evolving. Research regarding other bacterial species indicates a high frequency of mutation based resistance in conjunction with azithromycin use, i.e. when treating Mycoplasma genitalium infections. There has only been case reports of tetracycline resistance among human Chlamydia isolates, but a recent study suggest that there might be decreasing effectiveness also for doxycycline. Veterinaries has for several years observed increasing prevalence of tetracycline resistance among Chlamydia suis. Within the Chlamydia population there is promiscuous horizontal gene transfer.

If the current trend of declining cure rates continues, the investigators might face a situation where there are no documented and effective treatments for Chlamydia trachomatis infections. This underline an urgent need to expand the number of documented treatment options and mecillinam seems to be one of the options that warrant further investigation.

The objectives of this study is to prove the concept of treating genital Chlamydia trachomatis with mecillinam (Pivmecillinamhydrochlorid).

ELIGIBILITY:
Inclusion Criteria:

* Proficient in oral and written Norwegian
* Positive NAAT in first void urine for Chlamydia trachomatis
* Negative NAAT in first void urine for Mycoplasma genitalium
* Heterosexual male
* Asymptomatic

Exclusion Criteria:

* Known allergies for mecillinam, penicillin or cephalosporines
* Metabolic anomalies of aciduric type
* Apparent underweight
* Use of mecillinam within the last two months
* Under treatment with Valproat, other anti-infective drugs, immuno-modulating medication
* In the opinion of investigator,obvious reasons why patient will fails to adhere to treatment and follow-up protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Negative control test for Chlamydia in urine (NAAT; Nucleic Acid AmplificationTest) | 3 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Olaug Olsen, MD, PhD, Principal Investigator — Oslo UniversityHospital , Olafia Clinic
Locations (1):
- Olafia Clinic,Oslo University Hosptial, Oslo, Norway

REFERENCES:
- [Derived] Nilsen E, Aasterod M, Hustad PS, Olsen AO. Mecillinam against genital Chlamydia trachomatis infection: a small-scale proof-of-concept study shows a low cure rate. J Antimicrob Chemother. 2016 Aug;71(8):2270-2. doi: 10.1093/jac/dkw134. Epub 2016 May 10. PMID 27165786